CLINICAL TRIAL: NCT00314509
Title: ADVICE: A Dose Range Finding Study of Formoterol Administered Once Daily in the Evening in Combination With Ciclesonide Using the Ultrahaler™ Versus Monotherapy of Each Drug in Asthmatic Patients
Brief Title: Safety and Tolerability of Ciclesonide and Formoterol Fumarate Inhaled Once Daily in Patients With Asthma (18 to 75 y) (BY9010/M1-506)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BY9010/M1-506
Record Dates: First submitted 2006-04-11; First posted 2006-04-14 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Asthma
Keywords: Asthma; Ciclesonide; Formoterol Fumarate; Long-acting beta2-agonists; LABA; Steroids
MeSH Terms: conditions — Asthma | interventions — ciclesonide

INTERVENTIONS:
Drug: Ciclesonide/Formoterol Combination

SUMMARY:
The aim of the study is to compare the efficacy of two doses of a fixed combination of ciclesonide/formoterol fumarate versus ciclesonide alone versus formoterol fumarate alone in patients with asthma. The study duration consists of a baseline period (2 to 3 weeks) and a treatment period (8 weeks). The study will provide further data on safety and tolerability of ciclesonide/formoterol fumarate.

ELIGIBILITY:
Main Inclusion Criteria:

* Written informed consent
* Good health with the exception of bronchial asthma (for at least 6 months)
* FEV1 > 60% to < 80% of predicted (if pretreated with inhaled steroids only)
* FEV1 > 60% to ≤ 85% of predicted (if pretreated with inhaled steroids in combination with other asthma controller)

Main Exclusion Criteria:

* Concomitant severe diseases or diseases which are contraindications for the use of inhaled steroids or long-acting beta2-agonists
* Chronic obstructive pulmonary disease (COPD), i.e. chronic bronchitis or emphysema, and/or other relevant lung diseases causing alternating impairment in pulmonary function
* Current smoking or cessation of smoking within the last 6 months or previous smoking with a smoking history ≥ 10 cigarette pack-years
* Use of other drugs not allowed
* Pregnancy or intention to become pregnant during the course of the study, breast feeding, or lack of safe contraception in women of childbearing potential

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240
Dates: Start 2005-07; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Time to the first experience of lack of efficacy
AUC (FEV1) over a 24 h dosing interval.

SECONDARY OUTCOMES:
FEV1
morning and evening PEF, asthma symptoms and use of rescue medication
proportion of patients with a clinical asthma exacerbation.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (25):
- France (2):
  - Altana Pharma/Nycomed, Grenoble
  - Altana Pharma/Nycomed, Montpellier
- Germany (5):
  - Altana Pharma/Nycomed, Berlin
  - Altana Pharma/Nycomed, Großhansdorf
  - Altana Pharma/Nycomed, Mainz
  - Altana Pharma/Nycomed, Rüdersdorf
  - Altana Pharma/Nycomed, Wiesbaden
- Hungary (11):
  - Altana Pharma/Nycomed, Balassagyarmat
  - Altana Pharma/Nycomed, Balatonfüred
  - Altana Pharma/Nycomed, Budapest
  - Altana Pharma/Nycomed, Csorna
  - Altana Pharma/Nycomed, Debrecen
  - Altana Pharma/Nycomed, Győr
  - Altana Pharma/Nycomed, Mátraháza
  - Altana Pharma/Nycomed, Mosonmagyaróvár
  - Altana Pharma/Nycomed, Nyíregyháza
  - Altana Pharma/Nycomed, Szolnok
  - Altana Pharma/Nycomed, Szombathely
- South Africa (7):
  - Altana Pharma/Nycomed, Arcadia, Pretoria
  - Altana Pharma/Nycomed, Bellville, Cape Town
  - Altana Pharma/Nycomed, Bloemfontein
  - Altana Pharma/Nycomed, Cape Town, Tygerberg
  - Altana Pharma/Nycomed, Mowbray, Cape Town
  - Altana Pharma/Nycomed, Panorama / RSA-Cape Town
  - Altana Pharma/Nycomed, Pretoria

REFERENCES:
- See also: BY9010 M1-506.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4546&filename=BY9010%20M1-506.pdf